CLINICAL TRIAL: NCT06065917
Title: Set up and Validation of Total Small Bowel Length Measurement Using Computed Tomography and Magnetic Resonance Imaging With 3D Reconstruction and Artificial Intelligence Tool in Obese Patients Candidates to Metabolic Surgery
Brief Title: Total Small Bowel Length Measurement Using Computed Tomography and Magnetic Resonance Imaging in Obese Patients
Acronym: SBOM-AI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Collaborators: University of Padova (Other); Federico II University (Other)
Responsible Party: Principal Investigator, Niccolo Petrucciani, MD, PhD, Associate Professor of Surgery, University of Roma La Sapienza
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: C.88
Record Dates: First submitted 2023-09-13; First posted 2023-10-04 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Obesity; Bariatric Surgery Candidate
Keywords: obesity; artificial intelligence; computed tomography; bariatric surgery; small bowel lenght; metabolic surgery; magnetic resonance
MeSH Terms: conditions — Obesity | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Artificial intelligence training cohort and validation cohort (Experimental): Three high-volume Italian centers will enroll 195 obese patients who are candidates for metabolic surgery for obesity. Part of them will be established a training cohort (total = 105 patients), used to set up the AI-based method of TSBL measurement. The other 90 patients (30 for each center) will represent the validation cohort.
  Interventions: Diagnostic Test: Measurement of the total small bowel length using CT scan and MRI with 3D reconstruction and AI tool

INTERVENTIONS:
Diagnostic Test: Measurement of the total small bowel length using CT scan and MRI with 3D reconstruction and AI tool — The intervention consists in performing CT and MR imaging with small bowel length measurement before bariatric/metabolic surgery in obese patients. Then, during surgery the patients will undergo laparoscopic stretched small bowel measurement as the reference gold standard method to measure the small bowel length. The imaging of the training cohort will be used to trained an AI to set up an automatic method of small bowel length measurement via the analysis of CT and MRI imaging.

SUMMARY:
The aim of the study is to set up and validate a reliable and reproducible automated method using preoperative radiological imaging to measure the TSBL in patients undergoing laparoscopic bariatric/metabolic surgery.

DETAILED DESCRIPTION:
The total length of the small intestine (TSBL) represents a crucial parameter for obtaining a safe and successful minimally invasive surgery in metabolic/bariatric bypass surgery.

Nowadays, the standard of small intestine measurement is the intraoperative measurement. Laparoscopy represents the standard approach for baratric/metabolic, making the TSBL measurement time-consuming and risky in case of intestinal lesions. An accurate and effective non-invasive preoperative measurement of the TSBL will allow to evaluate the variability of the TSBL, which affects the surgical strategy. Cross-sectional imaging could play an important role in this setting thanks to the possibility of measuring in a non-invasive way the TSBL. Some studies performed with both Computed Tomography (CT) and Magnetic Resonance (MR) report promising results. However, they are limited by the small size of the sample, the lack of standardized technique and the lack of an automatic method based on Artificial Intelligence (AI).

The evaluation of a reliable preoperative method to measure TSBL using cross-sectional imaging will potentially reduce intraoperative complications and insufficient long-term weight loss or nutritional deficiencies. In this scenario a possible solution could be the implementation of analysis method through the development of an AI algorithm capable of automatically segmenting the small intestine.

The PRIMARY END POINT of this study is to set up and validate a reliable and reproductible automatic method to measure the TSBL in patients candidates for laparoscopic bariatric/metabolic surgery, based on preoperative radiological imaging

The main phases of the project will be:

1. evaluate the feasibility of preoperative CT and MRI-base measurement of the TSBL in a large cohort of obese patients and compare radiological measurement with intraoperative laparoscopic measurement (method of elongation) as a reference standard (1).
2. Evaluate the more accurate cross-sectional imaging between CT and MRI to measure the length of the small intestine.
3. Build an AI tool that can automatically measure TSBL on transversal slice imaging.

Three high-volume Italian centers will enroll 195 obese patients who are candidates for metabolic surgery for obesity. Part of them will be established training cohort (total = 105 patients), used to set up the AI-based method of TSBL measurement. The other 90 patients (30 for each center) will represent the validation cohort.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 35 kg/m2 and at least one obesity-related comorbidity
* BMI > 40 kg/m2
* failure of at least six months of dietary and/or medical treatment of obesity
* indication for intervention validated after multidisciplinary evaluation in a specific board meeting

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Estimated)
Dates: Start 2024-01-02 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Concordance between AI-based total small bowel length measure and laparoscopic total small bowel length measure | 1 month
  the main outcome is to set up and validate a reliable and reproducible automated method using preoperative radiological imaging to measure the TSBL in patients candidates for laparoscopic bariatric/metabolic surgery. The results of AI measurement will be compared with those of laparoscopic measurement to examine the level of concordance

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliera Universitaria Sant'Andrea, Rome, RM, Italy

IPD SHARING:
Plan to Share IPD: No